CLINICAL TRIAL: NCT04116528
Title: Opiate Suicide Study in Patients With Major Depression
Acronym: AFSP
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Stanford University (Other)
Responsible Party: Principal Investigator, Alan Schatzberg, Professor, Stanford University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 51536
Record Dates: First submitted 2019-07-03; First posted 2019-10-04 (Actual); Last update posted 2025-02-21 (Actual); Status verified 2025-02

CONDITIONS: Major Depressive Disorder
MeSH Terms: conditions — Depressive Disorder, Major | interventions — Ketamine; Buprenorphine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Ketamine (Other): Every eligible participant will receive 0.5mg/kg IV given over 40 minutes
  Interventions: Drug: Ketamine
- Buprenorphine or Placebo (Active Comparator): Buprenorphine or placebo once daily for 4 weeks
  Interventions: Drug: Buprenorphine; Drug: Placebo oral tablet

INTERVENTIONS:
Drug: Ketamine — 0.5mg/kg
  Arms: Ketamine
Drug: Buprenorphine — Buprenorphine (0.2-0.8mg/day) or Placebo orally dissolving tablet
  Arms: Buprenorphine or Placebo
Drug: Placebo oral tablet — Buprenorphine or Placebo orally dissolving tablet
  Arms: Buprenorphine or Placebo

SUMMARY:
To explore whether intravenous ketamine followed by buprenorphine produces more rapid and sustained anti-suicidal effects than ketamine followed by placebo, investigators will conduct a single study that will take approximately 2.5 years to complete. 60 subjects (60 infusions) or approximately 24 infusions per year.

DETAILED DESCRIPTION:
The investigators hypothesize that patients who receive buprenorphine following ketamine will demonstrate significantly greater anti-suicidal effects over the course of the study and maintained until four weeks of buprenorphine than will placebo. Buprenorphine subjects will also demonstrate longer times to recurrence than will those who receive ketamine followed by placebo. As secondary analyses, the investigators will test whether there is a relationship of improvement in sleep and pain to change in suicide ratings.

Aim 2: To assess the potential role played by the opioid properties of a single infusion of ketamine, investigators will for the ketamine portion determine ketamine and metabolite blood levels during and after the infusion as well as pupillary changes and correlate them to anti-suicidal response at Day 1. Investigators will also collect blood to determine buprenorphine blood levels, prolactin as well as collecting data on pupillary changes and then assess for potential relationships with anti-suicidal response.

ELIGIBILITY:
Inclusion Criteria:

* A subject will be eligible for inclusion only if all of the following criteria are met:

  1. Male or female, 18 to 70 years of age, inclusive, at screen.
  2. Able to read, understand, and provide written, dated informed consent prior to screening. Participants will be deemed likely to comply with study protocol and communicate with study personnel about adverse events and other clinically important information.
  3. Diagnosed with Major Depressive Disorder (MDD), single or recurrent or Bipolar-II Disorder and currently experiencing a Major Depressive Episode (MDE) of at least eight weeks in duration, prior to screening, according to the criteria defined in the Diagnosis and Statistical Manual of Mental Disorders, Fourth Edition, Text Revision(DSM-IV-TR™). The diagnosis of MDD will be made by a site psychiatrist and supported by the Structured Clinical Interview for DSM-IV-TR™ (SCID-I/P).
  4. Has a history of TRD during the current MDE, as assessed by the investigator. TRD is defined as failure to achieve a satisfactory response (e.g., less than 50% improvement of depression symptoms), as perceived by the participant, to at least one "treatment course" of a therapeutic dose of an antidepressant therapy of at least 8 weeks duration. The adequacy of dose and duration of the antidepressant therapy will be determined as per the MGH ATRQ criteria. Participants must currently be on a stable (for at least 4 weeks) and adequate (according to the MGH ATRQ) dose of ongoing SSRI or SNRI antidepressant therapy, of which total duration must be at least 8 weeks. Participants may also have a history of intolerance to at least 2 antidepressant medications. These patients with the intolerance history will not be required to be currently taking an antidepressant medication.
  5. Meet the threshold on the total SSI score of >/=6 at both screening and baseline visits.
  6. Participants must qualify as "Moderately Treatment Refractory" using the Maudsley staging method, which incorporates past treatments, severity of symptoms and duration of presenting episode.
  7. In good general health, as ascertained by medical history, physical examination (PE) (including measurement of supine and standing vital signs), clinical laboratory evaluations, and 3-lead electrocardiogram (ECG) if no evaluation available from the last 6 months.
  8. If female, a status of non-childbearing potential or use of an acceptable form of birth control per the following specific criteria:

     a. Non-childbearing potential (e.g., physiologically incapable of becoming pregnant, i.e., permanently sterilized (status post hysterectomy, bilateral tubal ligation), or is post-menopausal with her last menses at least one year prior to screening); or b. Childbearing potential, and meets the following criteria: i. Childbearing potential, including women using any form of hormonal birth control, on hormone replacement therapy started prior to 12 months of amenorrhea, using an intrauterine device (IUD), having a monogamous relationship with a partner who has had a vasectomy, or is sexually abstinent.

     ii. Negative urinary pregnancy test at screening, confirmed by a negative urinary pregnancy test at randomization prior to receiving study treatment.

     iii. Willing and able to continuously use one of the following methods of birth control during the course of the study, defined as those which result in a low failure rate (i.e., less than 1% per year) when used consistently and correctly: implants, injectable or patch hormonal contraception, oral contraceptives, IUD, double-barrier contraception, sexual abstinence. The form of birth control will be documented at screening and baseline.
  9. Body mass index between 17-40kg/m2.
  10. Concurrent psychotherapy will be allowed if the type (e.g., supportive, cognitive behavioral, insight-oriented, et al) and frequency (e.g., weekly or monthly) of the therapy has been stable for at least three months prior to screening and if the type and frequency of the therapy is expected to remain stable during the course of the subject's participation in the study.
  11. Concurrent hypnotic therapy (e.g., with zolpidem, zaleplon, melatonin, or trazodone) will be allowed if the therapy has been stable for at least 4 weeks prior to screening and if it is expected to remain stable during the course of the subject's participation in the study.

      Exclusion Criteria:
* A potential participant will NOT be eligible for participation in this study if any of the following criteria are met:

  1. Female of childbearing potential who is not willing to use one of the specified forms of birth control during the study.
  2. Female that is pregnant or breastfeeding.
  3. Female with a positive pregnancy test at screening or baseline.
  4. Total SSI score of <6 at the screen or baseline visits.

  6. Current diagnosis of a Substance Use Disorder (Abuse or Dependence, as defined by DSM-IV-TR™), with the exception of nicotine dependence, at screening or within six months prior to screening.

  7. Current diagnosis of Axis I disorders other than Dysthymic Disorder, Generalized Anxiety Disorder, Social Anxiety Disorder, Panic Disorder, Agoraphobia, or Specific Phobia (unless one of these is comorbid and clinically unstable, and/or the focus of the participant's treatment for the past six months or more).

  8. History of schizophrenia or schizoaffective disorders, or any history of psychotic symptoms in the current or previous depressive episodes.

  9. History of anorexia nervosa, bulimia nervosa, or eating disorder not otherwise specified, within one year of screening.

  10. Any Axis I or Axis II Disorder, which at screening is clinically predominant to their MDD or has been predominant to their MDD at any time within six months prior to screening. A diagnosis of borderline personality disorder is excluded.

  11. In the judgment of the investigator, the subject is at significant risk for suicidal behavior during the course of his/her participation in the study.

  12. Has dementia, delirium, amnestic, or any other cognitive disorder.

  13. Has a clinically significant abnormality on the screening physical examination that might affect safety, study participation, or confound interpretation of study results.

  14. Participation in any clinical trial with an investigational drug or device within the past month or concurrent to study participation.

  15. Known history or current episode of:
  1. QTcF (Fridericia-corrected) ≥450 msec at screening (Visit 1) or randomization
  2. Syncopal event within the past year.
  3. Congestive heart failure (CHF) New York Heart Association Criteria >Stage 2
  4. Angina pectoris
  5. Heart rate <50 or >105 beats per minute at screening or randomization

     16. Chronic lung disease.

     17. Lifetime history of surgical procedures involving the brain or meninges, encephalitis, meningitis, degenerative central nervous system disorder (e.g., Alzheimer's or Parkinson's Disease), epilepsy, mental retardation, or any other disease/procedure/accident/intervention associated with significant injury to or malfunction of the central nervous system (CNS), or a history of significant head trauma within the past two years.

     18. Presents with any of the following lab abnormalities w/in the past 6 months:

  <!-- -->

  1. Thyroid stimulating hormone (TSH) outside of the normal limits and clinically significant as determined by the investigator. Free thyroxine (T4) levels may be measured if TSH level is high. Subject will be excluded if T4 level is clinically significant.
  2. Any other clinically significant abnormal laboratory result at the time of the screening exam.

     19. History of hypothyroidism and has been on a stable dosage of thyroid replacement medication for less than six months prior to screening.(Subjects on a stable dosage of thyroid replacement medication for at least six months or more prior to screening are eligible for enrollment.)

     20. History of hyperthyroidism which was treated (medically or surgically) less than six months prior to screening.

     21. Any current or past history of any physical condition which in the investigator's opinion might put the subject at risk or interfere with study results interpretation.

     22. History of positive screening urine test for drugs of abuse at screening: cocaine, amphetamines, barbiturates, opiates.

     23. Current (or chronic) use of opiates. History of Opioid Use Disorder.

     24. Current use of lamotrigine and an inability to stop the medication prior to receiving ketamine.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2020-08-01 (Actual); Primary Completion 2025-04-28 (Estimated); Study Completion 2026-07-01 (Estimated)

PRIMARY OUTCOMES:
Change in Beck Suicidal Ideation Scale total scores will be analyzed as the primary outcome measure using analysis of variance model for repeated measures. | change from Day 3-31 and add to the model the Day 0 to 3 change in response to ketamine.
  The model will include the difference in total scores on the suicidality measure from days 3 to 31 as a within subject effect, treatment, and time, as well as time x treatment interaction. The model will include Day 3 score as well. The total scores range from 0 to 38, with higher values indicating a greater risk of suicide.All effects will use p<.05 for simple effects and p=0.1 for interactions, Using a sample size of 60, the hypothesis test will be fully powered (i.e., 80%) to detect effect sizes of 0.35 or greater.

SECONDARY OUTCOMES:
The investigators will assess opioid activity of ketamine as well as buprenorphine | Day 3-31
  peripherally by exploring opioid activity in subjects treated in the ketamine infusion and the sublingual buprenorphine vs. placebo phases by measuring serum metabolites of both ketamine and buprenorphine. The metabolites are measured in ng/mL with a reference interval of 1-10. Any presence of the drug will result in a number within the interval. If none detected, a not established level will be the result.

OTHER OUTCOMES:
Serum prolactin level | Day 1 and 3-31.
  Levels of the hormone prolactin may be increased by opioids and ketamine in serum.
Pupillometry | change from Day 3-31
  Moreover, we will apply pupillometry to estimate opioid activity. Levels of drug and opioid activity at specific time points will be correlated with response at that time point. In addition, regression analyses will be used to assess the relative contribution of opioid activity in blood, drug blood level, and pupil measure to improvement in suicidal behavior as well as mood, pain, and insomnia. This aim is exploratory.

CONTACTS AND LOCATIONS:
Overall Officials: Alan F. Schatzberg, Study Director — Stanford University
Locations (1):
- Stanford University School of Medicine, Stanford, California, United States